CLINICAL TRIAL: NCT00796939
Title: Randomized, Placebo-Controlled Trial of Short Wavelength Light Administered Just Prior to Waking in Young Men
Brief Title: Effects of Light Treatment During Sleep on Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Michael Grandner, PhD, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH068545 (NIH); R01MH068545 (NIH); MH68545; DATR A3-NSS
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Depression
Keywords: Delayed Sleep Phase Syndrome; Sleep
MeSH Terms: conditions — Depression; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green Light Mask (Active Comparator)
  Interventions: Device: Green light mask
- Red light mask (Placebo Comparator)
  Interventions: Device: Red Light Mask

INTERVENTIONS:
Device: Green light mask — Participants will receive approximately 10,000 lux from green light-emitting diodes.
  Arms: Green Light Mask
Device: Red Light Mask — Participants will receive approximately 0.5 lux from white light-emitting diodes covered by a red gel.
  Arms: Red light mask

SUMMARY:
This study will determine if green light exposure during sleep is effective in reducing mild depression symptoms in young men.

DETAILED DESCRIPTION:
The circadian rhythm is the human body's internal clock. It affects sleeping and wakefulness patterns. Some scientists theorize that a disruption of circadian rhythms, or other circadian abnormalities, can cause a depressed state. Light received through the eyes can alter the circadian rhythm, and sustained exposure to artificial bright light during the last half of usual sleep time can change the phase of the circadian rhythm. Several studies have found that exposure to bright white light in the morning hours is an effective treatment for depression, especially during the first week of depression treatment. Other studies have shown that green or blue light is preferable to yellow or red light in depression treatment. This study will expose young men to different types of light during the last part of their sleep cycle to determine whether the treatment is safe and tolerable and whether it reduces mood disturbance and depression. The study will also determine the light's effect on the production of luteinizing hormone (LH) and testosterone, hormones that may play a role in depression.

Participation in this study will last 15 days. At the beginning of the study, participants will be provided with study materials and instructed in their use. These materials will include a wrist actigraph, which is a sleep and wakefulness monitoring device similar to a wristwatch; a binder containing instructions, questionnaires, and forms; and a light mask. Participants will be randomly assigned to receive a light mask with either intense green or dim red light. Participants will wear the wrist actigraph throughout the study. For the first 3 days of the study, participants will sleep normally and fill out questionnaires and a sleep diary. The questionnaires will measure mood, sleepiness, sleep quality, treatment effects, and sleep time preference. The sleep diary will be a record of time spent sleeping, time it takes to fall asleep, number of times waking during the night, and similar measures. Starting on the third night, participants will wear the light mask when sleeping. Every day participants will fill out the questionnaires and sleep diary, and they will contact the study investigators to ensure compliance and to ask any questions. Participants will also provide saliva and urine samples once at the beginning and once at the end of the study. These samples will be used to test for testosterone and LH, respectively.

ELIGIBILITY:
Exclusion Criteria:

* Presence of clinical depression
* Presence of a sleep disorder

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Safety, measured through the Systematic Assessment for Treatment Emergent Effects (SAFTEE) questionnaire | Measured on Days 3 and 15
Tolerability, measured through compliance reports | Measured daily for the length of the study
Mood disturbance, measured on the Quick Inventory of Depressive Symptomology-Self Report (QIDS-SR) | Measured on Days 3 and 15

SECONDARY OUTCOMES:
Sleep diary | Measured daily for the duration of the study
Mood visual analog scale | Measured daily for the duration of the study
Luteinizing hormone, measured through urinalysis | Measured on Days 3 and 13
Testosterone, measured through saliva analysis | Measured on Days 3 and 13

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, La Jolla, California, United States